CLINICAL TRIAL: NCT02710006
Title: Feasibility and Reliability of Assessing Uterine Cavity Volume by SonoAVC in Women With Reproductive Failure.
Brief Title: Automatic Volume Calculations During Three-dimensional Sonohysterography.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwin & Ludwin Gynecology, Private Medical Center (Other)
Collaborators: Jagiellonian University (Other); University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Artur Ludwin, Artur Ludwin MD, PhD, Ludwin & Ludwin Gynecology, Private Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2/KBL/OIL/2016
Record Dates: First submitted 2016-03-06; First posted 2016-03-16 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Infertility,; Abortions, Spontaneous, Habitual
Keywords: Uterus; Ultrasound
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SonoHysteroAVC (Experimental): Three-dimensional sonohysterography is the first point for uterine cavity volume estimation, and it is going to be performed in all participants. The investigators are going to fill the uterine cavity twice by saline solution during single sonohysterography procedure, and acquise the volumetric datasets of uterus for offline analysis. The 3D dataset containing the entire uterine cavity will by analyzed using a personal computer and/or the ultrasound machine with specific softwere.
  Interventions: Procedure: Sonohysterography

INTERVENTIONS:
Procedure: Sonohysterography — Sonohysterography, also known as saline infusion sonography, is a special, minimally invasive ultrasound technique. Sonohysterography is a technique in which fluid is injected through the cervix into the uterus, and ultrasound is used to. It provides pictures of the inside of a woman's uterus. Three-dimensional sonohysterography is based on volumetric scanning of uterus and its cavity during saline infusion.
  Other Names: Saline infusion sonography

SUMMARY:
The purpose of this trial is to evaluate the feasibility and reliability of automatic volume calculation of uterine cavity in women with reproductive failures. 3D volumes of uterus and uterine cavity will be acquired during three-dimensional ultrasonography and sonohysterography. After that independent observers will measure offline the uterine cavity volume using automatic volume calculation using SonoAVC general software, and VOCAL software.

DETAILED DESCRIPTION:
INTRODUCTION

The uterus is one of key organs in reproduction and fetal development. A distorted shape and size of uterine cavity may to have significant impact on the reproductive failures (Chan et al., 2011; Saravelos et al., 2008). Current definitions and classification for uterine morphology and its congenital malformation are still controversial (Grimbizis et al., 2013; 2015; Ludwin and Ludwin, 2015a, b). This is an important barrier for studies evaluating the effectiveness of interventions for women with such conditions (Ludwin et al., 2015 a, b).

The uterine cavity volume is a specific feature of each individual uterus, and together with shape of uterine cavity may play one of the crucial roles in etiology of reproductive failures. To the investigators' knowledge the uterine cavity volume has never been studied in this context (Ludwin et al., 2016).

Recently, the technique of uterine cavity imaging, volume estimation, and quantification of deformity degree using automatic volume calculation (called SonoHysteroAVC; using SonoAVC software; GE Medical Systems, Zipf, Austria) during three-dimensional sonohysterography has been described (Ludwin et al., 2016). Uterine volume estimation is also potentially possible using Virtual Organ Computer-aided AnaLysis (VOCAL™; GE Medical Systems, Zipf, Austria), as for endometrial volume calculation (Martins et al., 2011).

The investigators believe that SonoHysteroAVC technique might improve the knowledge about uterine anatomy, the diagnostic accuracy of uterine cavity shape imaging, and the management of women with different morphological shapes of the uterine cavity. (Ludwin et al., 2016).

AIMS AND HYPOTHESES

Objective: to assess the inter-observer reliability of measuring the uterine cavity volume by automatic volume calculation.

Hypothesis: inter-observer reliability of the uterine cavity volume estimation using automatic volume calculation is very good.

Additional objective: to compare SonoAVC with VOCAL in uterine cavity volume estimation

DESIGN AND PATIENTS Design:Described elsewhere Setting:Described elsewhere Patients: Described elsewhere Inclusion criteria: Described elsewhere Exclusion criteria: Described elsewhere

Sample size:

The reliability estimates of uterine cavity automatic volume estimation are unknown. The feasibility of automatic volume calculation in deferent uterine condition also is unknown.

The investigators assumed that 100 subjects would be sufficient to obtain precise reliability coefficients (Streiner and Kottner, 2014), and 30 participants is minimal sample size for the feasibility study.

Interventions: Repeated three-dimensional sonohysterography (3D-SIS).

Data acquisition: two 3D data-sets of 3D-SIS per participant (observer 0; Obs0).

Analysis: Observer A (ObsA) will analyze the 1st data-set twice and the 2nd data-set once. Observer B (ObsB) will analyze the 2nd data-set once.

Comparisons:

ObsA-Dataset1 (1st analysis) vs. ObsA-Dataset1 (2nd analysis) to determine of repeatability ObsA-Dataset1 vs. ObsA-Dataset2 to determine variability caused by repeating the procedure ObsA-Dataset2 vs. ObsB-Dataset2 to determine inter-observer variability by reading ObsA-Dataset1 vs. ObsB-Dataset2 to determine inter-observer variability caused by repeating the exam

Outcomes:

i) The concordance correlation coefficient ii) Limits of agreement (LoA) iii) Time needed for acquisition iv) Time needed for analysis

Additional aim:

SonoAVC vs VOCAL (reproducibility and time needed)

Data processing and analysis: The researchers will ensure the confidentiality of sensitive data by minimizing the number of personnel who handles subject data.

Consent: All subjects will be given detailed explanation of the study and a written consent form will be signed by the patient and retained in the investigators' confidential records.

ELIGIBILITY:
Inclusion Criteria:

* infertility (12 months trying to conceive without success) and/or two previous miscarriages

Exclusion Criteria:

* unknown pregnancy (ultrasound examination)
* menopause
* precancerous conditions and cancers of female genital tract
* refused consent

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Concordance correlation coefficient in uterine cavity automated volume calculation | up to 12 months
  the concordance correlation coefficient measures the agreement between two variables to evaluate reliability
Limits of agreement (LoA) in uterine cavity volume estimation | up to 12 months
  Limits of agreement are an estimate of the interval within which a proportion of the differences between measurements lie.
Time needed for acquisition | up to 12 months
  Time needed for performing of three-dimensional sonohysterography and for uterine cavity 3D dataset acquisition (time of real-time three-dimensional sonohysterography)
Time needed for uterine cavity volume analysis | up to 12 months
  Time needed for performing of uterine cavity volume calculation in offline analysis

CONTACTS AND LOCATIONS:
Overall Officials: Artur Ludwin, MD, PhD, Principal Investigator — Ludwin & Ludwin Gynecology
Locations (1):
- Ludwin & Ludwin Gynecology, Specialist Medical Practice Artur Ludwin, Krakow, Malopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ludwin A, Ludwin I. Comparison of the ESHRE-ESGE and ASRM classifications of Mullerian duct anomalies in everyday practice. Hum Reprod. 2015 Mar;30(3):569-80. doi: 10.1093/humrep/deu344. Epub 2014 Dec 22. PMID 25534461
- [Background] Ludwin A, Ludwin I. Diagnostic rate and accuracy of the ESHRE-ESGE classification for septate uterus and other common uterine malformations: why do we not see that the Emperor is naked? Ultrasound Obstet Gynecol. 2015 Nov;46(5):634-6. doi: 10.1002/uog.14941. No abstract available. PMID 26525503
- [Background] Ludwin A, Ludwin I, Kudla M, Pitynski K, Banas T, Jach R, Knafel A. Diagnostic accuracy of three-dimensional sonohysterography compared with office hysteroscopy and its interrater/intrarater agreement in uterine cavity assessment after hysteroscopic metroplasty. Fertil Steril. 2014 May;101(5):1392-9. doi: 10.1016/j.fertnstert.2014.01.039. Epub 2014 Feb 26. PMID 24581576
- [Background] Martins WP, Raine-Fenning NJ, Leite SP, Ferriani RA, Nastri CO. A standardized measurement technique may improve the reliability of measurements of endometrial thickness and volume. Ultrasound Obstet Gynecol. 2011 Jul;38(1):107-15. doi: 10.1002/uog.9016. Epub 2011 Apr 28. PMID 21465609
- [Background] Coelho Neto MA, Roncato P, Nastri CO, Martins WP. True Reproducibility of UltraSound Techniques (TRUST): systematic review of reliability studies in obstetrics and gynecology. Ultrasound Obstet Gynecol. 2015 Jul;46(1):14-20. doi: 10.1002/uog.14654. Epub 2015 Jun 4. PMID 25175693
- [Background] Chan YY, Jayaprakasan K, Tan A, Thornton JG, Coomarasamy A, Raine-Fenning NJ. Reproductive outcomes in women with congenital uterine anomalies: a systematic review. Ultrasound Obstet Gynecol. 2011 Oct;38(4):371-82. doi: 10.1002/uog.10056. PMID 21830244
- [Background] Grimbizis GF, Gordts S, Di Spiezio Sardo A, Brucker S, De Angelis C, Gergolet M, Li TC, Tanos V, Brolmann H, Gianaroli L, Campo R. The ESHRE/ESGE consensus on the classification of female genital tract congenital anomalies. Hum Reprod. 2013 Aug;28(8):2032-44. doi: 10.1093/humrep/det098. Epub 2013 Jun 14. PMID 23771171
- [Background] Grimbizis GF, Di Spiezio Sardo A, Saravelos SH, Gordts S, Exacoustos C, Van Schoubroeck D, Bermejo C, Amso NN, Nargund G, Timmerman D, Athanasiadis A, Brucker S, De Angelis C, Gergolet M, Li TC, Tanos V, Tarlatzis B, Farquharson R, Gianaroli L, Campo R. The Thessaloniki ESHRE/ESGE consensus on diagnosis of female genital anomalies. Hum Reprod. 2016 Jan;31(1):2-7. doi: 10.1093/humrep/dev264. Epub 2015 Nov 4. PMID 26537921
- [Background] Ludwin A, Ludwin I, Kudla M, Kottner J. Reliability of the European Society of Human Reproduction and Embryology/European Society for Gynaecological Endoscopy and American Society for Reproductive Medicine classification systems for congenital uterine anomalies detected using three-dimensional ultrasonography. Fertil Steril. 2015 Sep;104(3):688-97.e8. doi: 10.1016/j.fertnstert.2015.06.019. Epub 2015 Jul 7. PMID 26158905
- [Background] Ludwin A, Martins WP, Ludwin I. Uterine cavity imaging, volume estimation and quantification of degree of deformity using automatic volume calculation: description of technique. Ultrasound Obstet Gynecol. 2017 Jul;50(1):138-140. doi: 10.1002/uog.15890. Epub 2017 May 28. No abstract available. PMID 26919726
- [Background] Streiner DL, Kottner J. Recommendations for reporting the results of studies of instrument and scale development and testing. J Adv Nurs. 2014 Sep;70(9):1970-1979. doi: 10.1111/jan.12402. Epub 2014 Mar 30. PMID 24684713